CLINICAL TRIAL: NCT01636713
Title: A 24-week Randomised, Double-blind and Placebo-controlled Study to Evaluate the Efficacy and Safety of GSK573719/GW642444 125/25 mcg and 62.5/25mcg Inhalation Powder Compared With Placebo Inhalation Powder Delivered Once-daily Via a Novel Dry Powder Inhaler in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 24-week Study to Evaluate the Efficacy and Safety of GSK573719/GW642444 125/25 mcg and 62.5/25mcg Inhalation Powder Compared With Placebo in Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114634
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK573719/VI 62.5/25 (Experimental): Inhalation via Novel Dry Powder Inhaler Once a day
  Interventions: Drug: GSK573719/VI 62.5/25
- GSK573719/VI 125/25 (Experimental): Inhalation via Novel Dry Powder Inhaler Once a day
  Interventions: Drug: GSK573719/VI 125/25
- Placebo (Placebo Comparator): Inhalation via Novel Dry Powder Inhaler Once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK573719/VI 62.5/25 — Inhalation via Novel Dry Powder Inhaler Once a day
  Arms: GSK573719/VI 62.5/25
Drug: GSK573719/VI 125/25 — Inhalation via Novel Dry Powder Inhaler Once a day
  Arms: GSK573719/VI 125/25
Drug: Placebo — Inhalation via Novel Dry Powder Inhaler Once a day
  Arms: Placebo

SUMMARY:
This is a 24-week, phase III multicenter, randomized, double-blind, placebo-controlled, parallel-group study. The study will have 9 scheduled visits and a telephone contact Follow-up visit one week following the end of study treatment.

The study primary endpoint is

-Clinic visit trough (pre-bronchodilator and pre-dose) FEV1 on Treatment Day 169 Trough FEV1 on Treatment Day 169 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Treatment Day 168 (i.e. at the Week 24 visit).

Secondary endpoints are;

* Mean TDI focal score at Week 24
* Weighted mean clinic visit FEV1 over 0 to 6 hours post-dose at Visit 2 (Day 1)

Eligible subjects will be randomised to GSK573719/GW642444 125/25mcg, GSK573719/GW642444 62.5/25mcg and placebo treatment groups in a 1:1:1 ratio such that of the planned 573 total number of randomised subjects, approximately 191 subjects will be randomised to each active treatment group and 191 subjects will be randomised to placebo. All treatments will be administered once daily in the morning by inhalation using a Novel Dry Powder Inhaler (NDPI).

There will be a total of 9 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit.1) will complete a 7 to 14 day Run-In period followed by a 24-week Treatment period. Clinic visits will be at screening, Randomisation (Day1), Day2, after 4, 8, 12, 16, and 24-weeks of treatment, and 1 day after the Week 24 Visit (also referred as Treatment Day 169). A Follow-Up contact for adverse event assessment will be conducted by telephone approximately 7 days after Visit 9 or the Early Withdrawal Visit. The total duration of subject participation, including Follow-up will be approximately 27 weeks. All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the Run-In and Study Treatment Periods.

At screening, pre-bronchodilator spirometry will be performed followed by post-albuterol/salbutamol spirometry testing. Post-albuterol/salbutamol FEV1 and FEV1/FVC values will be used to determine subject eligibility. To further characterise bronchodilator responsiveness, post ipratropium testing will be conducted following completion of post-albuterol/salbutamol spirometry.

Spirometry will be conducted at each post-randomisation clinic visit. Six hour post-dose serial spirometry will be conducted at Visit 2. Trough spirometry will be obtained 23 and 24 hours after the previous day's dose of blinded study medication at Visits 3 to 9.

Assessments of dyspnea will be obtained using the Baseline and Transition Dyspnoea Index (BDI/TDI) which is an interviewer based instrument. At Visit 2, the severity of dyspnoea at baseline will be assessed using the BDI. At subsequent visits (Visits 4, 6, and 8) change from baseline will be assessed using the TDI. Administration of the BDI and TDI should be done prior to spirometry and any other study-related procedures Disease specific health status will be evaluated using the St. George's Respiratory Questionnaire (SGRQ) and COPD Assessment Test (CAT), at baseline (Visit 2) and Visits 4, 6 and 8.

The occurrence of adverse events will be evaluated throughout the study beginning at Visit 2. SAEs will be collected over the same time period as for AEs. However, any SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded from the time a subject consents to participate in the study up to and including any follow up contact.

Vital signs (blood pressure and pulse rate), 12-lead ECGs and standard clinical laboratory tests (hematology and blood biochemistry) will be obtained at selected clinic visits.

For determination of subject disposition, subjects will be considered to have completed the study, upon completion of Visit 9. There is no plan to provide any of the active study treatments for compassionate use following study completion.

The Intent-to-Treat (ITT) population will be the primary population of interest, and is defined as all randomised subjects who have received at least one dose of the randomised study medication during the Treatment Period.

Supplementary study conduct information not mandated to be present in this protocol is provided in the accompanying Study Procedures Manual (SPM). The SPM will provide the site personnel with administrative and detailed technical information that does not impact subject safety.

ELIGIBILITY:
Inclusion Criteria:

1. Type of subject: outpatient.
2. Informed Consent: A signed and dated written informed consent prior to study participation.
3. Age: 40 years of age or older at Screening (Visit 1).
4. Gender: Male or female subjects are eligible to participate in the study.
5. COPD History: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society [Celli, 2004] as follows:
6. Tobacco Use and Smoking History: Current or former cigarette smokers with a history of cigarette smoking of more than or equal to 10 pack-years
7. Severity of Disease: A post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and a post-albuterol/salbutamol FEV1 of less than or equal to 70% of predicted normal values calculated using NHANES III reference equations at Visit 1 [Hankinson1999,Hankinson, 2010].
8. Dyspnea: A score of ≥2 on the Modified Medical Research Council Dyspnoea Scale (mMRC) at Screening (Visit 2)

Exclusion Criteria:

1. Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
2. Asthma: A current diagnosis of asthma.
3. Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis) and lung cancer are absolute exclusionary conditions. A subject, who in the opinion of the investigator has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant, bronchiectasis, pulmonary hypertension, sarcoidosis or interstitial lung disease.
4. Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for < 5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary).
5. Chest X-Ray: A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Visit 1 if a chest X-ray or CT scan is not available within 6 months prior to Visit 1.
6. Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
7. Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
8. Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
9. 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1, including the presence of a paced rhythm on a 12-lead electrocardiogram (ECG) which causes the underlying rhythm and ECG to be obscured. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility.
10. Screening Labs: Significantly abnormal finding from clinical chemistry and haematology tests at Visit 1.
11. Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
12. Medications prior to Screening: List are provided in the protocol
13. Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., less than 12 hours per day) is not exclusionary.
14. Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
15. Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
16. Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
17. Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- China (17):
  - GSK Investigational Site, Gaungzhou, Guangdong
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Zhanjiang, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Qingdao, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuxi
- Philippines (2):
  - GSK Investigational Site, Jaro, Iloilo City
  - GSK Investigational Site, Quezon City
- South Korea (4):
  - GSK Investigational Site, Gangdong-gu, Seoul
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
- Taiwan (6):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung Hsien
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Nan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met eligibility criteria at Screening (Visit 1) completed a 7 to 14-day run-in period and were then randomized to a 24-week treatment period.
Pre-assignment Details: A total of 739 participants were screened; 580 participants were randomized in a 1:1:1 ratio to receive either one of the active treatments or placebo. One participant was randomized but data was excluded from analysis as requested by the local Ethic Committee because the participant was not consented according to the GCP standards.
Groups:
- Placebo: Participants received matching placebo once daily (QD) via a dry powder inhaler (DPI) in the morning for 24 weeks.
- UMEC/VI 62.5/25 µg QD: Participants received umeclidinium bromide (UMEC)/vilanterol (VI) 62.5/25 micrograms (µg) QD via a DPI in the morning for 24 weeks.
- UMEC/VI 125/25 µg QD: Participants received UMEC/VI 125/25 µg QD via a DPI in the morning for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Started | 193 | 194 | 193
Completed | 161 | 166 | 170
Not Completed | 32 | 28 | 23
Not completed — Adverse Event | 16 | 16 | 7
Not completed — Lack of Efficacy | 6 | 6 | 2
Not completed — Protocol Violation | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4 | 8
Not completed — Met Protocol-defined Stopping Criteria | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD | Total
Number analyzed (Participants) | 193 | 194 | 193 | 580
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.78) | 64.0 (8.71) | 63.7 (8.26) | 64.0 (8.57)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 11 | 11 | 38
  Male | 177 | 183 | 182 | 542
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian-East Asian Heritage | 170 | 173 | 173 | 516
  Asian-South East Asian Heritage | 21 | 21 | 20 | 62
  Asian-Mixed Asian Heritage | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) on Day 169 (Week 24)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84, 112, 168, and 169. Baseline is defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Trough FEV1 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after the previous morning's dosing (ie., trough FEV1 on Day 169 is the mean of the FEV1 values obtained 23 and 24 hours after the morning dosing on Day 168). Change from Baseline at a particular visit was calculated as the trough FEV1at that visit minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline, smoking status, country/region, day, day by Baseline and day by treatment interactions. par.=participants.
Time Frame: Baseline and Day 169
Population: Intent-to-Treat (ITT) Population: all par. randomized to trt. who received at least one dose of randomized study drug. Par. represents those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 162 | 165 | 168
Liters | 1.040 (0.0147) | 1.191 (0.0146) | 1.256 (0.0146)
Statistical Analysis 1: Comparison: Placebo vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.151, 95% CI 2-sided [0.110 to 0.191] — Least squares mean difference=UMEC/VI 62.5/25 µg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.216, 95% CI 2-sided [0.175 to 0.257] — Least squares mean difference= UMEC/VI 125/25 µg minus Placebo

2. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Day 168 (Week 24)
Description: The TDI is an interviewer-administered instrument which measures the changes in the participant's dyspnea from Baseline. This questionnaire was collected on Days 28, 84 and 168. The scores in the TDI evaluate ratings for 3 different categories (functional impairment, magnitude of task in exertional capacity, and magnitude of effort). TDI scores ranged from -3 (major deterioration) to +3 (major improvement); total score = -9 to 9. Analysis was performed using a repeated measures model with covariates of treatment, Baseline dyspnea index (BDI) focal score, smoking status, country/region, day, day by Baseline dyspnea index (BDI) focal score and day by treatment interactions.
Time Frame: Day 168 (Week 24)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 162 | 162 | 168
Scores on a scale | 2.0 (0.20) | 2.7 (0.20) | 2.9 (0.20)

3. Secondary Outcome: Change From Baseline Weighted Mean (WM) 0-6 Hour FEV1 Obtained Post-dose at Day 1
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated using the 0-6-hour post-dose FEV1 measurements collected on Day 1, which included pre-dose (30 minutes [min] and 5 min prior to dosing) and post-dose at 15 min, 30 min, 1 hour, 3 hours, and 6 hours. Change from Baseline at Day 1was calculated as the WM at post -dose value on Day 1 minus Baseline (mean of the two assessments made 30 min and 5 min pre-dose on Day 1). Analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of treatment, Baseline FEV1 (mean of the two assessments made 30 and 5 minutes pre-dose on Day 1), smoking status, and country/region.
Time Frame: Baseline and Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 190 | 192 | 192
Liters | 0.015 (0.0075) | 0.174 (0.0075) | 0.197 (0.0075)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to 24 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for members of the ITT Population, comprising all participants randomized to treatment who received at least one dose of randomized study medication during the treatment period.
Arm/Group | Placebo | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Serious Adverse Events (participants affected / at risk) | 17/193 | 15/194 | 6/193
Other Adverse Events (participants affected / at risk) | 31/193 | 38/194 | 33/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=193) | UMEC/VI 62.5/25 µg QD (N=194) | UMEC/VI 125/25 µg QD (N=193)
Drowning (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 2
Septic shock (Infections and infestations) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 3
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of chronic (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=193) | UMEC/VI 62.5/25 µg QD (N=194) | UMEC/VI 125/25 µg QD (N=193)
Nasopharyngitis (Infections and infestations) | 18 | 17 | 18
Upper respiratory tract infection (Infections and infestations) | 11 | 19 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.